The impact of *Lepidium meyenii* (MACA) supplementation on basketball-related performance

and anti-fatigue ability: a double blind crossover study

Document Date: January 30, 2024

**Project summary** 

Supplementation with Lepidium meyenii (MACA) has been shown in animal studies to increase blood

lactate clearance and rapid lactate removal, which may be effective in reducing fatigue during

intermittent exercise. However, no studies have investigated the effects of MACA supplementation on

interval exercise and basketball performance. We hypothesized that MACA supplementation could

reduce fatigue and improve performance in elite healthy male basketball players. This study aimed to

determine the effectiveness of MACA compared to placebo on overall basketball performance. In this

randomized crossover study, ten elite healthy male basketball players were included. Following a

17:00 PM training routine, participants completed a two-week supplementation with 2000 mg of

MACA or placebo. After supplementation, participants underwent a Basketball Jump Shooting

Accuracy Test and Repeated Sprint Ability Test.

**General information** 

Protocol title: The impact of Lepidium meyenii (MACA) supplementation on basketball-related

performance and anti-fatigue ability: a double blind crossover study (Date: 30/01/2024; ID: NA)

1

**Funder:** This study was not funded by any organization.

#### INTRODUCTION.

1

2

3

4

5

6

7

8

9

10

11

12

13

14

15

16

17

18

19

Lepidium meyenii (MACA) is a Peruvian cruciferous vegetable growing more than 4000 m and cultivated for over 2000 years (1). Traditionally, the Andean people used MACA as food or medicine (2). They believed consumption of MACA improves stamina and strength (1). In the 13th century, Inca consumed MACA prior to entering battle to increase their energy (3). Now the MACA has attracted interest as a dietary supplement because of its potential positive effects on physical and sexual activity (4). Several studies have been conducted to examine its biological activity, and have shown increased endurance capacity and protection against exercise-induced oxidative stress (5-7). In animal experiments, supplementation with MACA was found to improve endurance exercise capacity and enhance clearance of metabolites such as blood lactate in mice (8-11). However, we found that most scientific research on the biological activity of MACA in humans has focused on improving sexual performance or fertility (12). To date, one study has demonstrated that 14 days of MACA supplementation improved 40km time trial performance and libido in trained male cyclists (7). Therefore, more well-designed, randomized, placebo-controlled studies are needed to assess the effect of MACA supplementation on the clearance of blood lactate and specific exercise performance. Basketball players perform a range of technical skills during the game, including speed, agility, anaerobic capacity, vertical jumping ability, and game-specific skills. This high-intensity interval exercise has been found to increase the accumulation of lactic acid in the blood and lead to induced fatigue (13-15). In animal studies, MACA supplementation has been demonstrated to increase the clearance of blood lactate (10, 16). However, no studies have examined the effects of MACA on basketball-related performance and lactate clearance in basketball players. We hypothesized that MACA supplementation could reduce fatigue and improve performance in trained healthy male basketball players, and aimed to determine the effectiveness of MACA compared to placebo in overall basketball performance.

## **METHODS**

# **Study Design**

The study used a double blind, randomized controlled, crossover, repeated measures, placebo (control) trial design. Participants were randomized on a 1:1 basis to supplement daily with MACA (MC)or placebo (PL) for two weeks before sport performance tests, and separated by 14 days. Randomization was performed using a permuted block design with a computer random number generator by a research assistant not involved in any other aspect of the study. All researchers and those involved in outcome assessments (i.e. basic data collection, individuals performing sport performance tests, data entry, and analyses) were blinded to group assignments. The study was approved by the Institutional Review Board of Jen-Ai Hospital - Dali Branch (JCH-IRB 111-24). Participants were informed of the risks and purposes of the study before written consent was obtained. The study

complied with the World Medical Association Declaration of Helsinki-Ethical Principles for Medical

Research Involving Human Participants. We adhered to the Consolidated Standards of Reporting Trials

(CONSORT) guidelines for reporting on randomized clinical trials (17).

# **Participants**

We recruited ten healthy male trained basketball players (age:  $20.1 \pm 0.3$  year; body mass:  $79.2 \pm 11.1$  kg; height:  $181.9 \pm 6.0$  cm; body fat:  $12.6 \pm 6.0\%$ ). The sample size computation was based on the study by Mark Stone (7). It revealed a significant improvement (p=0.01) in time to complete 40km from baseline to post supplementation in the MACA trial with only 8 subjects (7). All participants were college elite basketball players competing in a Taiwan university basketball association who voluntarily participated in this study. The inclusion criteria were: (i) healthy male adults, those individuals who are free of pain, insomnia, or other injuries recently, without any medication used in recent 2 months, (ii) basketball players competing in a Taiwan university basketball association for more than two years. Interested participants were excluded if they: (i) were below 20 years old, (ii) did not have won at least eighth place in national-level basketball competitions, (iii) were with cardiovascular diseases or any disease that made subjects feel ill. All exclusion criteria were determined by interview.

## **Study Setting**

All the study was conducted in the indoor basketball stadium at the National Taiwan University of

Sport. We control the temperature and humidity of the basketball stadium via the air conditioner. The

study commenced in June 2022 and supplementation and sport performance tests were completed in

September 2022.

## Protocol

60

61

62

63

64

65

66

67

68

69

70

71

72

73

74

75

76

77

# **Experimental procedure**

Participants completed a supplementation period of two weeks during which they were provided with 2000mg of either MACA (MacaPro@ Gelatinized Maca Powder, Lytone, Taipei, Taiwan) or a Placebo (100% corn-starch maltodextrin powder) after the daily training at 17:00 pm (7). The MACA supplement is derived from a concentrated 6:1 blend of black, red, and yellow MACA root compounds, with an 80:15:5 ratio respectively. The chemical composition of the MACA supplement, an extract consists of macamides as discussed in Zheng et al. (18). The plant name has been checked with "World Flora Online" (www.worldfloraonline.org). A ccording to the ingredient information of this product, no other ingredients are mentioned, it is a purified extract powder. This company is a major manufacturer of MACA. The main components of MACA have been analyzed by ultrahighperformance liquid chromatography (HPLC) (19). The MACA supplement or Placebo were supplied as orange-white capsules with the same appearance. After the supplement was given, the subject would be confirmed to have finished taking it. The subjects were asked to record the dietary status for three days since three days before each testing session to make sure the same diet was consumed, and educated the subjects to avoid eating or drinking irritating food and taking any form of health supplements or ergogenic agents until the end of the experiment, and ensured that ingesting the same diet and avoiding strenuous exercise on the day before the next experiment.

During the two weeks of the supplementation process, the subjects were asked about their usage status and physical condition every day. If they felt any discomfort or took other medications, they immediately stopped administering the supplements and then continued to observe and record the participants' physical condition and were excluded from the trial. They were replaced with different participants. All ten athletes completed the entire protocol without adverse events after MACA supplementation.

Three days before the test, we asked the participants to record their diet and to consume the same diet at the same time in the next experiment. On the day of the experiment, we used photographs to record the breakfast and lunch consumed by the participants and asked the participants to repeat the same meals in the second experiment. The nutritional composition of breakfast and lunch was  $11.9\pm2.4\%$  protein,  $41.6\pm16.7\%$  carbohydrate,  $26.8\pm6.1\%$  lipid, and  $1353.6\pm135.4$  kcal.

After two weeks of the supplement, participants begin formal experimentation after arriving at the basketball stadium at 15:00 p.m. First, the participants were asked to lie on a bench for 10 minutes with a heart rate monitor (Polar, Finland). After 10 minutes resting, the pre-exercise blood lactate level was collected by the nurses. The disposable pen needle was used for blood collection, and 75% alcohol was used to sterilize the puncture site and the fingertips.

They performed two identical warm-up exercises and three court-based fitness tests: (1) countermovement jump test, (2) Basketball Jump Shooting Accuracy Test and, (3) Interval sprint training. All outcome measures presented acceptable test-retest reliability (20-23). During the test, participants then provided ratings of perceived performance and perceived exertion (RPE) using 10-

point Likert scales (with 1 indicating a minimum response and 10 indicating a maximum response). Capillary blood samples were collected to assess the blood lactate concentration before and after the interval sprints test. All testing sessions were completed with a period of rest of at least 14 days for complete recovery and MACA wash-out.

## Countermovement jump test

The countermovement jump test is performed using GymAware (GymAware, Kinetic Performance Technology, Canberra, Australia) equipment (24). The participants first stands in front of the instrument with his feet shoulder-width apart, crosses his arms and squats down quickly until his thighs are parallel to the ground then immediately jumped upward as high as they could. Three jumps were measured with 1 minute rest for each participant. The mean height of the three jumps was obtained.

## **Basketball Jump Shooting Accuracy Test**

The first test was the basketball jump shooting Accuracy Test (BJSAT), which has been used in the past with sufficient reliability to two and three-point shooting accuracy (22). All athletes were given a demonstration and performed a 2-min shooting warm-up from the shot locations. They were instructed to attempt four shots with an even spread from the left and right sides of the court and from two- and three-point distance. In total, the test consisted of 8 x jump shot attempts at predetermined locations on the court. The shot order for the BJSAT ensured that athletes alternate between two-point

and three-point distances and do not take consecutive jump shots from either distance throughout the test. All shots were attempted with athletes placing both feet within a marked area at each shot location (60 cm x 60 cm). If an athlete attempted a jump shot with one or both feet outside of the marked area, the athlete continued the trial; however verbal instruction was given immediately to ensure both feet were placed within the marked area for the remaining shot attempts. The scoring methods is shown in Table 1. The male athletes used standard size 7 basketballs.

Table 1. Scoring criteria for the Basketball Jump Shooting Accuracy Test.

| Score | Description |
|-------|-------------------------------------------------------------------|
| 3 | The basketball passes through the basket without touching the rim |
| | or backboard. |
| 2 | The basketball make contact with the rim or backboard before |
| | passing through the basket. |
| 1 | The basketball makes contact with the rim or backboard, but does |
| | not pass through the basket. |
| 0 | The basketball does not come in contact with the rim or backboard |
| | and does not pass through the basket. |

# 

# **Repeated Sprint Ability Test**

After the 10 minutes rest and recovery, the participants perform the next test of Repeated Sprint Ability test (40× 15m with a 1:4, exercise: rest time ratio, such as 2 seconds: 8 seconds) (24). This test has been proven to reflect the sprinting ability of basketball players (25). Sprint direction was alternated for each sprint so the finish became the start for each consecutive sprint. There were several

types of repeat sprints test protocols. Half court, multiple change of direction protocol may not a typical repeat sprint test method, but it's a routine of their daily basketball training in Taiwan. Previous studies within the field have reported that familiarization is a crucial component as athletes typically find a preferable movement repertoire that enables them to achieve their best result (26).

## The lactate clearance rate

Between every 10 sprints, the participants walked back to the start point and rested. The capillary blood lactate, mean heart rate and RPE were measured after completion of each 10 times repeated sprint ability protocol. After full completion and resting in standing position for 5 minutes, the capillary blood lactate was taken and analyzed to measure the lactate clearance rate. The lactate clearance rate was calculated using the equation: Decreased percentage (%) = [(data during recovery period - data at exhaustion) / data at exhaustion ] × 100%. Finally, three vertical jump tests were measured after the whole test to be used as indicators of neuromuscular fatigue in the legs.

## **Statistical Analysis**

Data analysis was performed using SPSS software (version 20, Chicago, IL, USA). A descriptive analysis was performed using means and standard deviations. Normality of distribution was tested using the Shapiro-Wilk test. A two-way ANOVA Paired t-test was used to assess the differences in every 10 times repeated sprints, mean heart rate and RPE between MACA group and

placebo trials. Paired t-test was used to assess the differences in the Fatigue index, BJSAT score and
lactate clearance rate. The statistical power was s performed using G\*Power software package (Version
3.1.9.4, Kiel University). Statistical significance was set at p < 0.05.</li>

#### 156 References

- 157 1. Maca. LiverTox: Clinical and Research Information on Drug-Induced Liver Injury. Bethesda
- 158 (MD): National Institute of Diabetes and Digestive and Kidney Diseases; 2012.
- 159 2. Gonzales GF, Gonzales C, Gonzales-Castaneda C. Lepidium meyenii (Maca): a plant from the
- highlands of Peru–from tradition to science. Complementary Medicine Research. 2009;16(6):373-
- 161 80.
- 162 3. Hermann M. Andean roots and tubers: ahipa, arracacha, maca and yacon: International Potato
- 163 Center; 1997.
- 164 4. Gonzales GF, Gonzales C, Gonzales-Castañeda C. Lepidium meyenii (Maca): a plant from the
- highlands of Peru-from tradition to science. Forsch Komplementmed. 2009;16(6):373-80.
- 166 5. Tang W, Jin L, Xie L, Huang J, Wang N, Chu B, et al. Structural Characterization and Antifatigue
- 167 Effect In Vivo of Maca (Lepidium meyenii Walp) Polysaccharide. J Food Sci. 2017;82(3):757-64.
- 168 6. da Silva Leitão Peres N, Cabrera Parra Bortoluzzi L, Medeiros Marques LL, Formigoni M, Fuchs
- 169 RHB, Droval AA, et al. Medicinal effects of Peruvian maca (Lepidium meyenii): a review. Food Funct.
- 170 2020;11(1):83-92.
- 171 7. Stone M, Ibarra A, Roller M, Zangara A, Stevenson E. A pilot investigation into the effect of
- maca supplementation on physical activity and sexual desire in sportsmen. J Ethnopharmacol.
- 173 2009;126(3):574-6.
- 174 8. Zhu H, Xu W, Wang N, Jiang W, Cheng Y, Guo Y, et al. Anti-fatigue effect of Lepidium meyenii
- 175 Walp.(Maca) on preventing mitochondria-mediated muscle damage and oxidative stress in vivo and
- 176 vitro. Food & Function. 2021;12(7):3132-41.
- 177 9. Choi EH, Kang JI, Cho JY, Lee SH, Kim TS, Yeo IH, et al. Supplementation of standardized lipid-
- 178 soluble extract from maca (Lepidium meyenii) increases swimming endurance capacity in rats.
- 179 Journal of Functional Foods. 2012;4(2):568-73.
- 180 10. Tang W, Jin L, Xie L, Huang J, Wang N, Chu B, et al. Structural characterization and antifatigue
- 181 effect in vivo of maca (Lepidium meyenii Walp) polysaccharide. Journal of food science.
- 182 2017;82(3):757-64.
- 183 11. Li R-W, He J-C, Song D-H. Anti-physical fatigue effect of polysaccharides from Lepidium meyenii.
- 184 Walp. and the possible mechanisms. BIOMEDICAL RESEARCH-INDIA. 2017;28.
- 185 12. Lee MS, Lee HW, You S, Ha K-T. The use of maca (Lepidium meyenii) to improve semen quality:
- a systematic review. Maturitas. 2016;92:64-9.
- 187 13. McInnes SE, Carlson JS, Jones CJ, McKenna MJ. The physiological load imposed on basketball
- players during competition. J Sports Sci. 1995;13(5):387-97.
- 189 14. Stojanović E, Stojiljković N, Scanlan AT, Dalbo VJ, Berkelmans DM, Milanović Z. The Activity
- 190 Demands and Physiological Responses Encountered During Basketball Match-Play: A Systematic
- 191 Review. Sports Med. 2018;48(1):111-35.
- 192 15. Gottlieb R, Shalom A, Calleja-Gonzalez J. Physiology of Basketball–Field Tests. Review Article.
- 193 Journal of human kinetics. 2021;77(1):159-67.

- 194 16. Orhan C, Gencoglu H, Tuzcu M, Sahin N, Ojalvo SP, Sylla S, et al. Maca could improve endurance
- capacity possibly by increasing mitochondrial biogenesis pathways and antioxidant response in
- 196 exercised rats. J Food Biochem. 2022;46(7):e14159.
- 197 17. Schulz KF, Altman DG, Moher D. CONSORT 2010 statement: updated guidelines for reporting
- 198 parallel group randomised trials. Journal of Pharmacology and pharmacotherapeutics.
- 199 2010;1(2):100-7.
- 200 18. Zheng Y, Zhang WC, Wu ZY, Fu CX, Hui AL, Gao H, et al. Two macamide extracts relieve physical
- fatigue by attenuating muscle damage in mice. Journal of the Science of Food and Agriculture.
- 202 2019;99(3):1405-12.
- 203 19. McCollom MM, Villinski JR, McPhail KL, Craker LE, Gafner S. Analysis of macamides in samples
- of Maca (Lepidium meyenii) by HPLC-UV-MS/MS. Phytochemical Analysis: An International Journal
- of Plant Chemical and Biochemical Techniques. 2005;16(6):463-9.
- 206 20. Claudino JG, Cronin J, Mezêncio B, McMaster DT, McGuigan M, Tricoli V, et al. The
- 207 countermovement jump to monitor neuromuscular status: A meta-analysis. J Sci Med Sport.
- 208 2017;20(4):397-402.
- 209 21. Gathercole R, Sporer B, Stellingwerff T, Sleivert G. Alternative countermovement-jump analysis
- 210 to quantify acute neuromuscular fatigue. Int J Sports Physiol Perform. 2015;10(1):84-92.
- 21. Boddington BJ, Cripps AJ, Scanlan AT, Spiteri T. The validity and reliability of the Basketball
- Jump Shooting Accuracy Test. J Sports Sci. 2019;37(14):1648-54.
- 23. Paulauskas R, Kamarauskas P, Nekriošius R, Bigwood NM. Physical and Physiological Response
- 214 to Different Modes of Repeated Sprint Exercises in Basketball Players. J Hum Kinet. 2020;72:91-9.
- 215 24. Little T, Williams AG. Effects of sprint duration and exercise: rest ratio on repeated sprint
- 216 performance and physiological responses in professional soccer players. The Journal of Strength &
- 217 Conditioning Research. 2007;21(2):646-8.
- 218 25. Figueira B, Gonçalves B, Abade E, Paulauskas R, Masiulis N, Kamarauskas P, et al. Repeated
- 219 Sprint Ability in Elite Basketball Players: The Effects of 10 × 30 m Vs. 20 × 15 m Exercise Protocols on
- 220 Physiological Variables and Sprint Performance. J Hum Kinet. 2021;77:181-9.
- 221 26. Sekulic D, Spasic M, Mirkov D, Cavar M, Sattler T. Gender-specific influences of balance, speed,
- and power on agility performance. The Journal of Strength & Conditioning Research.
- 223 2013;27(3):802-11.

224

225